CLINICAL TRIAL: NCT05273411
Title: The Effect of Different Ketone Supplements on Blood Beta-hydroxybutyrate (β-OHB) and Blood Glucose in Healthy Individuals
Brief Title: The Effect of Different Ketone Supplements on β-OHB and Blood Glucose in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Dr. Jonathan Little, Associate Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: H22-00083
Record Dates: First submitted 2022-03-01; First posted 2022-03-10 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-02

CONDITIONS: Ketosis; Blood Glucose
MeSH Terms: conditions — Ketosis | interventions — 3-Hydroxybutyric Acid; 1,3-butylene glycol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester (Active Comparator): 1 x 20 mL
  Interventions: Dietary Supplement: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester
- Beta-hydroxybutyric acid (Experimental): 1 x 237 mL
  Interventions: Dietary Supplement: Beta-hydroxybutyric acid
- 1,3-Butanediol (Experimental): 1 x 35 mL
  Interventions: Dietary Supplement: 1,3-Butanediol

INTERVENTIONS:
Dietary Supplement: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester — Single-dose pharmacokinetic study over 4 hours.
  Other Names: Exogenous Ketones
  Arms: (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester
Dietary Supplement: Beta-hydroxybutyric acid — Beta-hydroxybutyric acid
  Other Names: Exogenous Ketones
  Arms: Beta-hydroxybutyric acid
Dietary Supplement: 1,3-Butanediol — 1,3-Butanediol
  Other Names: Exogenous Ketones
  Arms: 1,3-Butanediol

SUMMARY:
Ketone bodies are a fuel source and signaling molecule that are produced by your body during prolonged fasting or if you consistently eat at low-carbohydrate diet. Blood ketones can be used as a source of energy during fasting and are used by your brain as an alternative source of fuel to glucose. Previous studies have found that ketones, when consumed in form of a supplement drink, can increase blood ketone levels and lower blood glucose, the amount of sugar in your blood. This is of potential interest for individuals with high blood sugar, such as people living with type 2 diabetes. However, there are different types of ketone supplements that differ in how they are metabolized in the body. Little is known about how these supplements affect blood ketone and blood glucose levels. The main objective of this study is to determine the effect of three different ketone supplements on blood ketones and blood glucose. The results of this pilot study will be used to guide future research for larger and more extensive studies on ketone supplements.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18;
* able to fast overnight

Exclusion Criteria:

* being a competitive endurance athlete;
* following a ketogenic diet, low-calorie diet, periodic fasting regimen, or regularly consuming ketogenic supplements;
* being unable to travel to and from the university;
* being unable to follow the diet instructions;
* being pregnant or planning to become pregnant during the study;
* having been diagnosed with a chronic disorder of glucose or fat metabolism, including type 2 diabetes, chronic pancreatitis, or gallbladder disease;
* being unable to read or communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2022-05-18 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The investigators will share individual patient data (de-identified) with researchers upon request.

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: 1 x 20 mL; (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester; single-dose pharmacokinetic study over 4 hours.
  1 x 237 mL; Beta-hydroxybutyric acid; single-dose pharmacokinetic study over 4 hours.
  1 x 35 mL; 1,3-Butanediol; single-dose pharmacokinetic study over 4 hours.
- Arm 2: 1 x 20 mL; (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester; single-dose pharmacokinetic study over 4 hours.
  1 x 35 mL; 1,3-Butanediol; single-dose pharmacokinetic study over 4 hours.
  1 x 237 mL; Beta-hydroxybutyric acid; single-dose pharmacokinetic study over 4 hours.
- Arm 3: 1 x 35 mL; 1,3-Butanediol; single-dose pharmacokinetic study over 4 hours.
  1 x 237 mL; Beta-hydroxybutyric acid; single-dose pharmacokinetic study over 4 hours.
  1 x 20 mL; (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester; single-dose pharmacokinetic study over 4 hours.
- Arm 4: 1 x 35 mL; 1,3-Butanediol; single-dose pharmacokinetic study over 4 hours.
  1 x 20 mL; (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester; single-dose pharmacokinetic study over 4 hours.
  1 x 237 mL; Beta-hydroxybutyric acid; single-dose pharmacokinetic study over 4 hours.
- Arm 5: 1 x 237 mL; Beta-hydroxybutyric acid; single-dose pharmacokinetic study over 4 hours.
  1 x 35 mL; 1,3-Butanediol; single-dose pharmacokinetic study over 4 hours.
  1 x 20 mL; (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester; single-dose pharmacokinetic study over 4 hours.
- Arm 6: 1 x 237 mL; Beta-hydroxybutyric acid; single-dose pharmacokinetic study over 4 hours.
  1 x 20 mL; (R)-3-hydroxybutyl (R)-3-hydroxybutyrate ketone monoester; single-dose pharmacokinetic study over 4 hours.
  1 x 35 mL; 1,3-Butanediol; single-dose pharmacokinetic study over 4 hours.
Period: Intervention Period 1
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 2
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention Period 3
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Arm 4 | Arm 5 | Arm 6
Started | 2 | 2 | 2 | 2 | 2 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Single-dose pharmacokinetic study over 4 hours, three-way crossover study of three different ketone supplements (see description).
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 12

OUTCOME MEASURES:

1. Primary Outcome: Blood Beta-hydroxybutyrate
Description: Are under the curve (AUC) across 240 minutes after supplement consumption (assessed at baseline and 15, 30, 60, 90, 120, 180, and 240 post-supplementation)
Time Frame: 240 minutes (assessed at baseline and 15, 30, 60, 90, 120, 180, 240 minutes post-supplementation)
Measure: Mean (Standard Deviation); unit: area under the curve (mmol/L x 240 min)
Arm/Group | (R)-3-hydroxybutyl (R)-3-hydroxybutyrate Ketone Monoester | Beta-hydroxybutyric Acid | 1,3-Butanediol
Number analyzed (Participants) | 12 | 12 | 12
area under the curve (mmol/L x 240 min) | 217 (51) | 192 (63) | 176 (59)

2. Secondary Outcome: Blood Glucose
Description: Area under the curve (AUC)
Time Frame: 240 minutes (assessed at baseline and 15, 30, 60, 90, 120, 180, 240 minutes post-supplementation)
Reporting Status: Not Posted

3. Secondary Outcome: Blood Pressure
Description: Change over time
Time Frame: 240 minutes (assessed at baseline and 15, 30, 60, 90, 120, 180, 240 minutes post-supplementation)
Reporting Status: Not Posted

4. Secondary Outcome: Heart Rate
Description: Change over time
Time Frame: 240 minutes (assessed at baseline and 15, 30, 60, 90, 120, 180, 240 minutes post-supplementation)
Reporting Status: Not Posted

5. Secondary Outcome: Supplement Acceptability & Taste
Description: Questionnaire
Time Frame: 240 minutes post-supplementation
Reporting Status: Not Posted

6. Secondary Outcome: Hunger & Fullness
Description: Questionnaire
Time Frame: 240 minutes post-supplementation
Reporting Status: Not Posted

7. Secondary Outcome: Gastrointestinal Discomfort
Description: Questionnaire
Time Frame: 60 minutes post-supplementation
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Over the course of the three acute in-laboratory testing days
Description: Adverse events were any events reported or experienced by participants. We did not assess all-cause mortality as this was an acute one-day study.
Arm/Group | (R)-3-hydroxybutyl (R)-3-hydroxybutyrate Ketone Monoester | Beta-hydroxybutyric Acid | 1,3-Butanediol
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT05273411/Prot_SAP_000.pdf